CLINICAL TRIAL: NCT05529082
Title: The Attitudes and Beliefs of Hispanic/Latino Individuals Toward Prescription Opioids and Non-Medical Opioid Use
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutional of Health (Unknown); UT Health Science Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-0543; NCI-2022-06839 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Opioids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Opioid Attitudes and Beliefs survey: Participants will complete a questionnaire about your feelings/beliefs on prescription pain medication and your experience with opioids/pain medication. Demographic information about you (such as your age, gender, race, ethnicity, and so on) will also be collected.
  Interventions: Other: Opioid Attitudes; Other: Beliefs survey

INTERVENTIONS:
Other: Opioid Attitudes — Participants will complete a questionnaire about your feelings/beliefs on prescription pain medication and your experience with opioids/pain medication. Demographic information about you (such as your age, gender, race, ethnicity, and so on) will also be collected.
Other: Beliefs survey — Participants will complete a questionnaire about your feelings/beliefs on prescription pain medication and your experience with opioids/pain medication. Demographic information about you (such as your age, gender, race, ethnicity, and so on) will also be collected.

SUMMARY:
To better understand how people think and feel about prescribed pain medication, including opioids.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objectives:

1. To examine the general attitudes and beliefs of Hispanic/Latino individuals about the use of prescription opioids. The primary outcomes include the responses to questions 13-28 from the Opioid Attitudes and Beliefs survey.

Secondary

1. To evaluate Hispanic/Latino individuals' reports of personal experiences with the use of opioids. The corresponding outcomes are the responses to questions 1-12 from the Opioid Attitudes and Beliefs survey.
2. To find out any potential reasons why some Hispanic/Latino individuals may refuse to use clinically indicated opioid prescriptions. These outcomes are the responses to questions 14-15 from the Opioid Attitudes and Beliefs survey.
3. To explore factors associated with participant's comfort with the use opioid analgesics for their pain. The outcome will be the association between participants' responses to question 2 and their characteristics such as age, gender, race, level of education, extent of acculturation, knowledge of opioids, or previous opioid use.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 years or older.
2. Ability to understand, read, write, or speak English and/or Spanish.
3. Ability to give informed consent.
4. Willingness to participate in the survey.

Exclusion criteria:

1. Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Opioid Attitudes and Beliefs Survey | through completion of study an average of 1 year
  The survey questionnaire consists of a total of 33 items in five brief sections and responses are mainly based on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Arthur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org